CLINICAL TRIAL: NCT05293522
Title: A Phase 2a, Multicenter, Randomized, Subject and Evaluator Blinded, Controlled Study Evaluating the Safety and Efficacy of NTX-001 Compared to Standard of Care in the Treatment and Prevention of Facial Paralysis Requiring Surgical Repair.
Brief Title: A Study of NTX-001 in the Treatment and Prevention of Facial Paralysis Requiring Surgical Repair.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment Rate
Sponsor: Neuraptive Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTx21202
Record Dates: First submitted 2022-02-14; First posted 2022-03-24 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-09

CONDITIONS: Facial Paralysis
Keywords: Parotidectomy; Nerve Transfers; Free functional muscle flaps
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NTX-001 (Experimental): Solution #1, Solution #2 Active, Solution #3
  Interventions: Combination Product: NTX-001
- Standard of Care (No Intervention): Standard neurorrhaphy

INTERVENTIONS:
Combination Product: NTX-001 — 2 solutions plus a delivery device; one time use surgical product
  Arms: NTX-001

SUMMARY:
This study involves the use of an Investigational Product called NTX-001. It is a product used in the repair of nerve injuries. It is used in the operating room. The main purposes of this study are to 1) see how safe NTX-001 is when used in nerve repair and, 2) see if your nerve becomes functional in a shorter period of time when compared to what is normally done to treat nerve injuries.

DETAILED DESCRIPTION:
Facial paralysis can be a consequence of traumatic facial nerve injury, iatrogenic causes, malignancy, congenital syndromes, and viral infections. Prolonged paralysis can result in ocular complications, articulation difficulties, impaired feeding, and difficulty in conveying emotion through expressive movement. The current treatment for permanent facial paralysis is facial reanimation surgery, which encompasses a broad range of procedures that restore form and function to the paralyzed face.

The importance of understanding the health utility of facial paralysis and the value of facial reanimation surgery increases. PEG-fusion is a promising therapy for patients that have or will have nerve conditions or injuries resulting in facial palsy that can be addressed surgically. Patients that have clinical evidence of facial paralysis requiring facial nerve repair from conditions or interventions that have or may result in paralysis will be evaluated for participation. The primary objective is to assess the safety of NTX-001 across 12 months following the nerve repair. The study will measure improvement in Facial Grading System (FG) for efficacy. Additionally, measures will include an EMG evaluation for assessment of nerve function intraoperatively, image-based automatic facial landmark analysis, improvement in Facial Clinimetric Evaluation Scale score, and Patient Global Impression of Change Response (PGIC).

ELIGIBILITY:
Inclusion Criteria:

The subject has clinical evidence of facial paralysis requiring facial nerve repair from conditions or interventions that have or may result in paralysis.

Exclusion Criteria:

Subjects whose nerve repair will occur greater than 48 hours after nerve transection.

Subjects requiring repair of the intracranial portion of the facial nerve. Subjects requiring repair involving an allograft or conduit except for procedures that require grafting of the other nerve branches when repairing the main facial nerve.

Subjects with Bell's palsy that have signs of spontaneous recovery by 12 months.

Subjects who, in the judgment of the investigator, are not likely to demonstrate meaningful recovery within 6 weeks due to significant facial muscle atrophy.

Subjects on chronic corticosteroid therapy within 14 days of repair.

The subject has documented history or clinical signs of:

Clinically significant neuropathy from any cause i.e., medications, chemotherapy, diabetes; Clinically significant systemic neuromuscular disease; Clinically significant local or systemic neurological deficit from other than the condition under study such as stroke; Or other treatments are known to affect the growth and/or physiology of the neural and vascular system with the exception of radiation therapy; The subject has a known allergy to polyethylene glycol (PEG) or human-grade silicone.

The subject is not able to strictly adhere to the rules of the current clinical protocol, e.g., significant mental health issues, homelessness, incarceration, intellectually or developmentally challenged without proper legal representation.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events for Safety | Adverse events will be assessed and recorded from start of study through 48 weeks or approximately 1 year..
  Measuring the safety of NTX-001 following the nerve repair based on the number of reported adverse events.
Sunnybrook Facial Grading System | From screening visit, and at weeks 6, 12, 24, 36, and 48.
  Change in Sunnybrook Facial Grading score from baseline as compared to Week 6;

OTHER OUTCOMES:
Intraoperative EMG | Once in the operating room.
  Electromyography (EMG) measures amplitude and duration of facial motor unit action potentials which reflects in the number of innervated muscle fibers. This may demonstrate if reinnervation or nerve conduction has been restored in the operating room.
Image-based automatic facial landmark identification system | From screening visit, and at weeks 1, 6, 12, 24, 36, and 48.
  Image analysis automatically identifies facial landmarks and uses the position of those landmarks to estimate facial symmetry and/or evaluate facial neuromuscular diseases.
Facial Clinimetric Evaluation Scale | From screening visit, and at weeks 6, 12, 24, 36, and 48.
  FaCE is a patient questionnaire that measures the patient's perception of their facial movement, facial comfort, oral function, eye comfort, tear control, and social function. Each one is scored separately to a total of 100, where 0 is the worst possible score to 100 is the best.
Patient Global Impression of Change | From screening visit, and at weeks 6, 12, 24, 36, and 48.
  PGIC is a patient questionnaire that evaluates the patients perception of their overall health status. A single-question with answers on a 7-point scale scored as: (1) "very much better," (2) "much better," (3) "a little better," (4) "no change," (5) "a little worse," (6) "much worse," or (7) "very much worse." The following ranges demonstrate disease worsening (0-3 points), stable disease (4 points) or disease improvement (5-7 points) since the initial baseline or prior assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Schulman, MD, Study Director — Chief Medical Officer
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - University of Indiana, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No